CLINICAL TRIAL: NCT06260592
Title: The Effect of the Level of Ethical Attitude Towards Care on the Skills of Humanistic Acting in Intensive Care Nurses
Brief Title: Ethical Attitude and Humanistic Acting Skills of Intensive Care Nurses
Status: Completed | Type: Observational
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Sponsor
Other Study IDs: Aysun Acun 4
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-02

CONDITIONS: Humanistic Care Skills
Keywords: nursing; Humanistic Care; intensive care nursing; ethic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- intensive care nurses: Ethical compliance and humanistic care of intensive care nurses.

SUMMARY:
Today, rapidly developing technology and changing treatment and care conditions increase the tendency towards ethical values both as an intellectual concept and as a moral guide. The nursing profession, which focuses on people in ethical terms, is also performed by people. This situation brings with it many ethical dilemmas in areas where health care services are provided. In ICUs, long and critical treatments of patients, differences of opinion between the medical team and the institution, non-compliance with patient rights, difficulties in terminal patient care, procedures performed without the patient's consent, distribution of limited medical resources, unethical attitudes and attitudes of nurse colleagues, Many issues such as long-term exposure to stressors and constant alarm sounds can cause mental distress and negative emotions in intensive care nurses. One of the effective ways to increase the quality of care provided by nurses is humanistic practice ability. The presence of humanistic practice ability provides more realistic, human-centered nursing care, improves the quality of life of patients, and also positively affects health expenditures.

DETAILED DESCRIPTION:
One of the effective ways to increase the quality of care provided by nurses is humanistic practice ability. The presence of humanistic practice ability provides more realistic, human-centered nursing care, improves the quality of life of patients, and also positively affects health expenditures. The humanist approach is increasing its importance day by day in planning individual care, evaluating the outcomes of care practices, and health-promoting information programs. In this context, it is of great importance to develop the humanist practice skills, humanist nursing spirit, humanist clinical practices and humanist nursing education of nurses who are actively involved in ICUs, as in all areas of care practice. In developing nurses' humanistic nursing behaviors, their level of knowledge and behavioral skills should first be revealed.

When the literature was examined, it was seen that there were studies examining the extent to which nurses experienced ethical problems and dilemmas during caregiving, their attitudes, and ethical decision-making processes. While studies on nurses' ethical decision-making processes are important, it is thought that studies measuring their level of humanistic behavior will also contribute to nursing care. This research aims to show the effect of intensive care nurses' ethical attitude levels on their ability to act humanistically. The research is original in that it combines ethical attitudes and humanistic behavior. It is anticipated that the research will contribute to nursing care and the knowledge base of the nursing profession.

ELIGIBILITY:
Inclusion Criteria:

* Becoming an intensive care nurse
* Volunteering to participate in the study

Exclusion Criteria:

* Not being an intensive care nurse
* Not volunteering to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nurses actively involved in the intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Ethical compliance of nurses in the intensive care unit | 06/02/2024-20/02/2024

SECONDARY OUTCOMES:
Humanistic care skills of nurses in the intensive care unit | 06/02/2024-20/02/2024

CONTACTS AND LOCATIONS:
Locations (1):
- Bilecik Şeyh Edebali University, Bilecik, Turkey (Türkiye)